CLINICAL TRIAL: NCT02412072
Title: Comparison of Dilatation & Curettage and Endometrial Aspiration Biopsy Accuracy in Patients Treated With Progestin for Endometrial Hyperplasia: A Korean Gynecologic Oncology Group Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korean Gynecologic Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: kgog2019
Record Dates: First submitted 2015-04-04; First posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Endometrial Hyperplasia
Keywords: Endometrial hyperplasia; Progesterone; LNG-IUS; dilatation & curettage; endometrial aspiration sampling
MeSH Terms: conditions — Endometrial Hyperplasia; Dilatation, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective multicenter trial has been started in Korea to evaluate the diagnostic accuracy of endometrial aspiration biopsy compared with D&C in patients treated with progestin for endometrial hyperplasia (EH). For conservative treatment of EH, oral progestins are most commonly used method with various treatment regimens and more recently, the levonorgestrel-releasing intrauterine system (LNG-IUS) also has been used successfully to treat EH. However, there is no report about the accuracy of endometrial sampling during hormonal treatment for follow-up evaluation of EH. Patients with histologically confirmed EH are offered hormonal treatment, one of the following 3 options: oral medroxyprogesterone acetate(MPA) 10mg/day for 14days per cycle, continuous oral MPA 10mg/day, or insertion of LNG-IUS. Histological surveillance is performed at 3-months or 6-months following initial treatment. Endometrial tissues are obtained via endometrial aspiration biopsy using a pipelle and D&C. In case of using LNG-IUS, endometrial aspiration biopsy will be done with LNG-IUS in uterus and then, after removal of LNG-IUS, D&C will be done. The biopsy findings will be compared. The primary endpoint is the consistency of the results of the endometrial aspiration biopsy and D&C. The secondary endpoint is the response rate with 3 types of progestin treatment at 6 months.

DETAILED DESCRIPTION:
Endometrial hyperplasia (EH) is a premalignant lesion of endometrial cancer (EC), which is the most common gynecological malignancy in developed countries [1]. Therefore, accurate diagnostics and proper management of EH are clinically significant to prevent EC development.

The treatment modality of EH mostly depends on the histological diagnosis and the woman's desire to retain fertility. The risk of cancer progression is low for women with non-atypical EH (<5%) but increases up to 30% for women with atypical EH [2, 3]. In this respect, hysterectomy is recommended for the treatment of atypical EH. Meanwhile, for patients with non-atypical EH or for young patients with atypical EH who strongly desire to preserve their fertility, various conservative therapies using progestin have been used. Traditionally, orally administered progestins such as megestrol acetate (MA) and medroxyprogesterone acetate (MPA) are most commonly used method with various treatment regimens [4, 5]. More recently, the levonorgestrel-releasing intrauterine system (LNG-IUS), which achieves higher local concentrations of progestogens in the endometrium, with lower systemic side effects, also has been used successfully to treat EH [6-12].

However, there is no report about the accuracy of endometrial sampling during hormonal treatment for EH or the best technique for follow-up evaluation of EH. A recent study comparing the histological results of pipelle biopsy and D&C reported almost equal EH-diagnostic success rates [13]. Meanwhile, these results were obtained for cases where the LNG-IUS was not in the uterus and where there were no progestin effects on the endometrium.

Therefore, the investigators conducted a large multicenter prospective study to compare the diagnostic accuracy of endometrial aspiration biopsy with dilatation & curettage (D&C) in follow up evaluation of patients treated with progestin for EH.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are histological confirmed as endometrial hyperplasia
2. Patients who desire to preserve fertility potential.
3. Patients signed the written informed consent voluntarily.

Exclusion Criteria:

1. Pregnancy or suspected pregnancy.
2. Patients who have severe underlying disease or complication.
3. Treatment for metastatic cancer from other organs or cancer therapy within the preceding 5 years.
4. Congenital or acquired uterine anomaly, including fibroids if they distort the uterine cavity.
5. Acute liver disease or kidney disease
6. Thrombosis or phlebothrombosis requiring treatment.
7. Genital (vaginal, uterine or ovarian) infection.
8. Acute severe disease of the arteries, such as stroke or heart infarction, or a history of artery disease.
9. Hypersensitivity to any component of this product.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with biopsy proven endometrial hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
consistency of the endometrial aspiration biopsy and D&C after hormonal treatment of EH | 3months or 6 months

SECONDARY OUTCOMES:
response rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam CAH medical center, Seoul, Gangnamgu, South Korea

REFERENCES:
- [Derived] Kim MK, Seong SJ, Park DC, Hong JH, Roh JW, Kang SB. Comparison of diagnostic accuracy between endometrial curettage and aspiration biopsy in patients treated with progestin for endometrial hyperplasia: a Korean Gynecologic Oncology Group study. J Gynecol Oncol. 2020 Jul;31(4):e51. doi: 10.3802/jgo.2020.31.e51. Epub 2020 Feb 7. PMID 32266800